CLINICAL TRIAL: NCT00635609
Title: Randomized, Open-label Study to Evaluate the Efficacy and Safety of Doryx Tablets Compared to Doxycycline Hyclate in the Treatment of Acne Vulgaris.
Brief Title: Treatment of Acne Vulgaris With Doryx Tablets Compared to Doxycyline Hyclate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-08607
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline hyclate (Doryx) (Experimental)
  Interventions: Drug: Doxycycline hyclate (Doryx)
- Doxycycline hyclate (Active Comparator)
  Interventions: Drug: Doxycycline hyclate

INTERVENTIONS:
Drug: Doxycycline hyclate (Doryx) — 150mg/day, oral, delayed release tablets
  Other Names: Doryx
  Arms: Doxycycline hyclate (Doryx)
Drug: Doxycycline hyclate — 100 mg/day, oral, tablets, immediate release
  Arms: Doxycycline hyclate

SUMMARY:
Randomized, multi-center, open label, active-comparator study to compare the efficacy and tolerability of Doryx Delayed Release Tablets to doxycycline hyclate in patients with moderate to severe acne vulgaris.

DETAILED DESCRIPTION:
Efficacy of Doryx Delayed Release Tablets to doxycycline hyclate will be assessed using an Investigator's Global Assessment (IGA) score and the absolute change from baseline to 12 weeks in inflammatory lesion count in patients with moderate to severe facial acne vulgaris. Additionally, the absolute change from baseline to 12 weeks in non-inflammatory lesions count of Doryx Delayed Release Tablets compared to doxycycline hyclate will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Must be 12 years of age or older.
* Has a diagnosis of facial acne vulgaris with no more than two nodules on the face.

Exclusion Criteria:

* Is allergic to tetracycline-class antibiotics or to any ingredient in the study medication.
* Has a history of pseudomembranous colitis or antibiotic-associated colitis.
* Has a history of hepatitis or liver damage or renal impairment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Secci, MD, Study Director — Warner Chilcott
Locations (4):
- United States (4):
  - Warner Chilcott Investigational Site, Vista, California
  - Warner Chilcott Investigational Site, Miami, Florida
  - Warner Chilcott Investigational Site, Louisville, Kentucky
  - Warner Chilcott Investigational Site, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxycycline Hyclate (Doryx) Delayed-release Tablets: Doxycycline hyclate (Doryx) delayed-release tablets, 150 mg once daily
- Doxycycline Hyclate Immediate-release Tablets: Doxycycline hyclate immediate-release tablets, 100 mg once daily
Period: Overall Study
Arm/Group | Doxycycline Hyclate (Doryx) Delayed-release Tablets | Doxycycline Hyclate Immediate-release Tablets
Started | 48 | 45
Completed | 41 | 42
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline Hyclate (Doryx) Delayed-release Tablets | Doxycycline Hyclate Immediate-release Tablets | Total
Number analyzed (Participants) | 48 | 45 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 21 | 49
  Between 18 and 65 years | 20 | 24 | 44
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 19.3 (5.8) | 20.9 (7.9) | 20.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 31 | 29 | 60
Region of Enrollment [Number; unit: participants]
  United States | 48 | 45 | 93
Ethnic Origin [Number; unit: participants]
  Hispanic | 27 | 26 | 53
  Not of Hispanic origin | 21 | 19 | 40
Race [Number; unit: participants]
  Asian or Pacific Islander | 0 | 1 | 1
  Black | 3 | 5 | 8
  Caucasian | 22 | 18 | 40
  Other | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Successful Outcome According to Investigator's Global Assessment (IGA)
Description: The Investigator's Global Assessment (IGA) was performed at baseline and at 12 weeks. The IGA score is based on a 5-point acne severity scale from zero (clear) to 4 (severe). Successful outcome is at least a 2-point reduction in IGA score from baseline to 12 weeks.
Time Frame: baseline and 12 weeks
Measure: Number; unit: participants
Arm/Group | Doxycycline Hyclate (Doryx) Delayed-release Tablets | Doxycycline Hyclate Immediate-release Tablets
Number analyzed (Participants) | 48 | 45
participants | 18 | 19
Statistical Analysis 1: Comparison: Doxycycline Hyclate (Doryx) Delayed-release Tablets vs Doxycycline Hyclate Immediate-release Tablets; Study not adequately powered to detect differences in efficacy outcomes. Results to provide estimates of safety and efficacy outcomes; Test type: Superiority or Other; p = 0.765, Cochran-Mantel-Haenszel; Stratified on investigational site

2. Secondary Outcome: Change From Baseline in Non-inflammatory Acne Lesion Count on the Face at 12 Weeks
Description: Acne lesions fall into 2 groups: inflammatory and non-inflammatory. The number of non-inflammatory acne lesions on the face was measured at baseline and after 12 weeks. The difference (change) was calculated.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Acne lesion count
Arm/Group | Doxycycline Hyclate (Doryx) Delayed-release Tablets | Doxycycline Hyclate Immediate-release Tablets
Number analyzed (Participants) | 48 | 45
Acne lesion count | 23.2 (19.3) | 27.6 (20.0)
Statistical Analysis 1: Comparison: Doxycycline Hyclate (Doryx) Delayed-release Tablets vs Doxycycline Hyclate Immediate-release Tablets; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.290, Cochran-Mantel-Haenszel; Stratified on investigational site

3. Primary Outcome: Change From Baseline in Inflammatory Acne Lesion Count on the Face at 12 Weeks
Description: Acne lesions fall into 2 groups: inflammatory and non-inflammatory. The number of inflammatory acne lesions on the face was measured at baseline and after 12 weeks. The difference (change) was calculated.
Time Frame: baseline and 12 weeks
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: acne lesion count
Arm/Group | Doxycycline Hyclate (Doryx) Delayed-release Tablets | Doxycycline Hyclate Immediate-release Tablets
Number analyzed (Participants) | 48 | 45
acne lesion count | 21.8 (13.8) | 26.6 (12.5)
Statistical Analysis 1: Comparison: Doxycycline Hyclate (Doryx) Delayed-release Tablets vs Doxycycline Hyclate Immediate-release Tablets; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.033, Cochran-Mantel-Haenszel; Stratified on investigational site

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Doxycycline Hyclate (Doryx) Delayed-release Tablets | Doxycycline Hyclate Immediate-release Tablets
Serious Adverse Events (participants affected / at risk) | 1/48 | 1/45
Other Adverse Events (participants affected / at risk) | 10/48 | 11/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline Hyclate (Doryx) Delayed-release Tablets (N=48) | Doxycycline Hyclate Immediate-release Tablets (N=45)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) — Intensity severe, unlikely related
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Intensity severe, unlikely related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline Hyclate (Doryx) Delayed-release Tablets (N=48) | Doxycycline Hyclate Immediate-release Tablets (N=45)
Headache (Nervous system disorders) | 7 (7) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Sunburn (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less